CLINICAL TRIAL: NCT01003171
Title: An Open-Label, Multiple-Dose Study of MCS-2 to Examine the Pharmacokinetics of MCS and Other Components After Once-daily Oral Dosing in Healthy Adult Volunteers
Brief Title: Pharmacokinetics of MCS in Healthy Volunteers
Acronym: MCS-2-US-pk
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Health Ever Bio-Tech Co., Ltd. (Industry)
Responsible Party: Fu-Feng Kuo / General Manager, Health Ever Bio-Tech Co., Ltd.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCS-2-US-pk
Record Dates: First submitted 2009-10-26; First posted 2009-10-28 (Estimated); Last update posted 2011-06-30 (Estimated); Status verified 2011-06

CONDITIONS: Healthy
Keywords: Pharmacokinetics; PK; MCS; Benign Prostatic Hyperplasia; Multi-Carotenoids; Healthy subjects
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MCS-2 (Experimental)
  Interventions: Drug: MCS-2 soft-gel capsule

INTERVENTIONS:
Drug: MCS-2 soft-gel capsule — MCS-2 30 mg/day
  Other Names: MUS

SUMMARY:
This study is to examine the pharmacokinetics, absorption and serum concentrations of MCS and other components after once-daily oral dosing of MCS.

DETAILED DESCRIPTION:
This study is an open-label, multiple-dose study, whose objective is to examine the pharmacokinetics of MCS and other components after once-daily oral dosing for 21 days.

Subjects will undergo a 14-day washout phase and then enter the 21-day treatment phase. During the treatment phase, subjects will receive MCS, once-daily within one hour after the evening meal. After completion of the treatment phase, subjects will enter a post-treatment 42-day washout phase. Throughout each of these phases, blood samples will be collected and assayed for concentrations of MCS and other components. The duration of protocol participation is expected to be 77 days for each eligible subject who completes the study.

ELIGIBILITY:
Inclusion Criteria:

* Normal healthy volunteers
* 18 years of age or older

Exclusion Criteria:

* Subjects who can not comply with the study procedures or sign the informed consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2011-08; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Serum MCS and other components levels | 21 days

SECONDARY OUTCOMES:
Incidence of treatment-emergent adverse events | 21 days